CLINICAL TRIAL: NCT04951986
Title: Testing New Strategies for Patients Hospitalised With HIV-associated Disseminated Tuberculosis
Acronym: NEW-STRAT TB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Charlotte Schutz, Co-Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC REF: 001/2021
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Disseminated Tuberculosis; HIV
Keywords: HIV; High dose rifampicin; Fluoroquinolones; Glucocorticoids; Antiretroviral therapy
MeSH Terms: interventions — Rifampin; Levofloxacin; Pyrazinamide; Ethambutol; Isoniazid; Prednisone

STUDY DESIGN:
Intervention Model Description: First intervention (open label):
  a) Experimental arm: Standard first-line anti-tuberculosis therapy plus additional rifampicin to reach 35mg/kg/day for 14 days plus levofloxacin 750mg/day for weight <50kg and 1g/day for weight >50kg for 14 days b) Control arm: Standard TB therapy containing rifampicin 10mg/kg for 14 days (standard of care) After 14 days both study arms will continue standard TB therapy with rifampicin at 10mg/kg to complete 2 months of intensive phase in total. This will be followed by standard continuation phase TB therapy.
  2. Second intervention (double-blind):
  1. Experimental arm: Prednisone 1.5mg/kg per day for 14 days
  2. Control arm: Identical placebo for 14 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose Rifampicin plus Levofloxacin (Experimental): Standard TB treatment plus additional Rifampicin 35 mg/kg/day PLUS Levofloxacin for 14 days
  Interventions: Drug: Rifampin; Drug: Levofloxacin; Drug: Rifampicin, Pyrazinamide, Ethambutol and Isoniazid
- Prednisone (Experimental): Prednisone 1.5 mg/kg for 14 days
  Interventions: Drug: Prednisone
- Standard TB treatment (Active Comparator): High dose rifampicin/levofloxacin comparator
  Interventions: Drug: Rifampicin, Pyrazinamide, Ethambutol and Isoniazid
- Placebo (Placebo Comparator): Prednisone comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifampin — Rifampicin up to 35 mg/kg/day for 14 days
  Other Names: rifampicin; Rifadin; Rimactane
  Arms: High dose Rifampicin plus Levofloxacin
Drug: Levofloxacin — Levofloxacin 750mg daily (for weight <50kg) or 1 g daily (for weight >50 kg) daily for 14 days
  Arms: High dose Rifampicin plus Levofloxacin
Drug: Rifampicin, Pyrazinamide, Ethambutol and Isoniazid — Rifampicin 10 mg/kg; Isoniazid 5 mg/kg; Pyrazinamide 15 mg/kg; Ethambutol15 mg/kg in fixed dose combination administered per weight band. Standard of care control arm
  Other Names: Rifafour
  Arms: High dose Rifampicin plus Levofloxacin; Standard TB treatment
Drug: Prednisone — Prednisone 1.5mg/kg/day for 14 days
  Other Names: Trolic
  Arms: Prednisone
Drug: Placebo — Placebo identical to Prednisone
  Arms: Placebo

SUMMARY:
The New Strat-TB trial is a superiority Phase III randomised control clinical trial with a 2X2 factorial design. The main aim of the study is to assess the efficacy and safety of high dose rifampicin and levofloxacin for 14 days in addition to standard TB therapy with or without steroids among adults hospitalized with HIV-associated disseminated tuberculosis.

The investigators hypothesize that intensified treatment with increased rifampicin doses at 35 mg/kg plus levofloxacin will more rapidly reduce the mycobacterial load. The investigators also hypothesize that steroids will have an immune-modulatory effect and dampen the activation of the innate immune system. The investigators hypothesize that these two strategies will lead to improved survival in patients hospitalized with HIV-associated disseminated tuberculosis.

DETAILED DESCRIPTION:
Primary efficacy endpoint:

All-cause mortality at 12 weeks

Secondary efficacy endpoint:

All-cause mortality at 2 and 24 weeks

Safety and tolerability endpoints:

* Occurrence of hepatotoxicity using the American Thoracic Society (ATS) hepatotoxicity criteria: Alanine aminotransferase (ALT) elevation of more than three times the upper limit of normal (ULN) in the presence of hepatitis symptoms and/or jaundice or five times the upper limit of normal in the absence of symptoms.
* Corticosteroid-associated adverse events, classified by severity and relation to study drug and will be reported if these develop within 4 weeks of enrolment. These will include new hypertension, new poor blood pressure control in a known hypertensive, hyperglycaemia, hypomania, mania, depression, acne, gastritis symptoms, upper gastrointestinal bleeding, and avascular bone necrosis.
* Laboratory safety data (Grade 3 and 4 abnormalities using the ACTG grading system): liver function tests (alanine and aspartate aminotransferase[ALT, AST], gammaglutamyl transferase [GGT], alkaline phosphatase [ALP], International Normalized Ratio [INR], conjugated and total bilirubin [CBR, TBR]), glucose, full blood counts (including white cell, neutrophil and platelet counts plus haemoglobin) and electrolytes (sodium, potassium) and creatinine.
* Occurrence of other opportunistic infections (AIDS-related, bacterial, fungal and viral) and malignancies (Kaposi's sarcoma) up to 12 weeks.
* Occurrence of paradoxical tuberculosis immune reconstitution inflammatory syndrome (TB-IRIS) in patients starting antiretroviral therapy up to 12 weeks.
* All grade 3 and 4 clinical adverse events (using the ACTG grading system)
* Serious adverse events
* Adverse events requiring study drug interruption and or withdrawal
* Adverse drug reactions attributed to study drug

Follow-up:

Participants will be followed up daily while admitted to hospital for assessment of adverse events. Safety and routine blood tests will be done on day 2, 4, 7, 14 and 28. Further visits will be on week 12 and 24.

Data monitoring:

The trial will be monitored by an independent Data and Safety Monitoring Board (DSMB) comprising 4 independent researchers and an independent statistician. If there is evidence of harm related to study medication or trial conduct the DSMB may advise the sponsor that trial enrolment should be stopped.

Clinical trial site:

Mitchells Plain Hospital and Khayelitsha Hospital

ELIGIBILITY:
Inclusion Criteria:

* Aged >18
* HIV infection
* Disseminated TB confirmed by one or more of the following tests being positive

  1. Lysed blood Xpert Ultra positive for MTB
  2. Concentrated urine Xpert Ultra positive for MTB
  3. Urine Alere LAM positive
* Hospital clinical team made decision to initiate TB treatment

Exclusion Criteria:

* Pregnant or breastfeeding
* Active or recent SARS-CoV-2 infection
* TB treatment within the last 1 month or more than 2 doses of TB treatment
* Rifampicin resistance
* Neurological TB
* Receiving corticosteroids or other immunosuppressive therapy
* ALT >120 IU/L or total bilirubin >34 μmol/L
* Plasma CrAg positive or cryptococcal meningitis
* Current malignancy requiring active treatment (including any Kaposi sarcoma lesions)
* Patients established on ART with Protease Inhibitor based regimen who cannot be switched to a dolutegravir based regimen
* Diabetic ketoacidosis or Hyperosmolar Non-ketotic acidosis
* Any condition in the opinion of the investigator for which participation would increase risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 weeks

SECONDARY OUTCOMES:
In-hospital mortality during index admission | 7 days
All-cause mortality | 2 and 24 weeks respectively

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Khayelitsha Hospital, c/o Steve Biko and Walter Sisulu Drives, Khayelitsha, Cape Town, Western Cape
  - Mitchells Plain Hospital, Mitchells PLain, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on request, after discussion with ethics committee
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Namale PE, Boloko L, Vermeulen M, Haigh KA, Bagula F, Maseko A, Sossen B, Lee-Jones S, Msomi Y, McIlleron H, Mnguni AT, Crede T, Szymanski P, Naude J, Ebrahim S, Vallie Y, Moosa MS, Bandeker I, Hoosain S, Nicol MP, Samodien N, Centner C, Dowling W, Denti P, Gumedze F, Little F, Parker A, Price B, Schietekat D, Simmons B, Hill A, Wilkinson RJ, Oliphant I, Hlungulu S, Apolisi I, Toleni M, Asare Z, Mpalali MK, Boshoff E, Prinsloo D, Lakay F, Bekiswa A, Jackson A, Barnes A, Johnson R, Wasserman S, Maartens G, Barr D, Schutz C, Meintjes G. Testing novel strategies for patients hospitalised with HIV-associated disseminated tuberculosis (NewStrat-TB): protocol for a randomised controlled trial. Trials. 2024 May 8;25(1):311. doi: 10.1186/s13063-024-08119-4. PMID 38720383

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT04951986/SAP_000.pdf